CLINICAL TRIAL: NCT01953055
Title: Phase II Study of Stereotactic Ablative Radiotherapy Including Regional Lymph Node Irradiation for Patients With High Risk Prostate Cancer (SATURN)
Brief Title: SABR Including Regional Lymph Node Irradiation for Patients With High Risk Prostate Cancer (SATURN)
Acronym: SATURN
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Andrew Loblaw, Dr. Andrew Loblaw, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALOB-SATURN2013
Record Dates: First submitted 2013-09-25; First posted 2013-09-30 (Estimated); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Prostate Cancer
Keywords: stereotactic ablative radiotherapy; androgen deprivation therapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stereotactic ablative radiotherapy (Experimental): 40 Gy in 5 fractions over 4 weeks to prostate; 25 Gy in 5 fractions over 4 weeks to pelvic lymph nodes given simulataneously.
  Interventions: Radiation: Stereotactic ablative radiotherapy

INTERVENTIONS:
Radiation: Stereotactic ablative radiotherapy

SUMMARY:
Current treatment options for high risk localized prostate cancer include radical prostatectomy +/- postoperative radiotherapy, radical radiotherapy with androgen deprivation therapy. Evidence has emerged that prostate cancer has a low α/β ratio in the range of 1-3 Gy. Even with high risk tumors, prostate cancer is hypothesized to have a greater sensitivity to large fraction sizes and high dose per fraction radiotherapy theoretically allows for biological dose escalation with fewer visits and no additional toxicity. Therefore, we hope to determine the toxicity, quality of life, biochemical and pathological control of SBRT for high risk prostate cancer incorporating ENI.

ELIGIBILITY:
Inclusion Criteria:

* informed consent obtained
* men > 18 years of age
* histologically confirmed prostate adenocarcinoma (centrally reviewed)
* high risk prostate cancer, defined as at least one of clinical stage T3 or Gleason 8-10, or PSA > 20ng/mL

Exclusion Criteria:

* prior pelvic radiotherapy
* anticoagulation medication (if unsafe to discontinue for gold seed insertion)
* diagnosis of bleeding diathesis
* large prostate (>90cm3) on imaging at time of gold seed insertion
* no evidence of castrate resistance (defined as PSA < 3ng/mL while testosterone is < 0.7nmol/L
* definitive regional or distant metastatic disease on staging investigations

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-11 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Acute GU and GI toxicities | Baseline to 3 months post treatment
  Acute GU and GI toxicities as assessed using the Common Terminology for Adverse Events (CTCAE) v3.0

SECONDARY OUTCOMES:
Late GU and GI toxicities | > 6 months post treatment
  Late GU and GI toxicities as assessed using RTOG grading schema
Quality of Life (QoL) | 5 years
  Quality of life using the Expanded Prostate Cancer Index Composite (EPIC) questionnaire
Biochemical control | 5 years
  Biochemical disease free survival
Disease free survival | 2 years
  Prostate biopsy 2 years post ADT cessation

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Loblaw, MD, Principal Investigator — Sunnybrook Health Sciences Centre/University of Toronto
Locations (1):
- Odette Cancer Centre/Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada